CLINICAL TRIAL: NCT02996396
Title: Multicenter, Observational, Registry to Assess Outcomes of Patients Treated With the CE Marked Nellix® System for Endovascular Abdominal Aortic Aneurysm Repair"
Brief Title: Nellix Registry Study: EVAS-Global
Acronym: EVAS FORWARD 2
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Endologix (Industry)
Responsible Party: Sponsor
Other Study IDs: CP0010 Ver. 2
Record Dates: First submitted 2016-12-12; First posted 2016-12-19 (Estimated); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: AAA, Aortoiliac Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients diagnosed with AAA who are considered candidates for Endovascular Repair and meet the study eligibility criteria and sign the Informed consent may be subsequently enrolled in the study.
  Interventions: Device: Nellix Endovascular Aneurysm Sealing System (Nellix®-System)

INTERVENTIONS:
Device: Nellix Endovascular Aneurysm Sealing System (Nellix®-System) — The Nellix system is comprised of two independent flow channels, one to each iliac artery. Each flow channel consists of a balloon-expanded ePTFE covered stent surrounded by a Polymer-filled EndoBag which fills the blood lumen within the aorta, and seals the aneurysm from side-branch flow.
  Other Names: Nellix EVAS FORWARD 2

SUMMARY:
Multicenter, single arm, open label, registry study with consecutive, eligible patient enrollment at each site. All subjects undergoing the Endovascular Aneurysm Sealing System (EVAS) with the Nellix®-System. Subjects will be followed procedurally to discharge, and as per institutional standard of care thereafter through to 5 years (total follow-up commitment)

ELIGIBILITY:
Inclusion Criteria:

1. Male or female at least 18 years old
2. Subject has signed informed consent for data release
3. Subjects with with AAA and eligible for endovascular repair

Exclusion Criteria:

1. Currently participating in another study where primary endpoint has not been reached yet
2. Known allergy to any of the device components
3. Pregnant (females of childbearing potential only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with AAA who are considered candidates for Endovascular Repair and meet the study eligibility criteria and sign the Informed consent may be subsequently enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2023-11-21 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with Immediate Procedural Technical Success | 30 Days
  Technical success is defined as successful delivery and deployment of the Nellix System in the planned location.
Safety assessment by Number of subjects with absence of Major Adverse Events (MAEs) | 30 Days
  Safety endpoint is measured with the number of subjects who are reported freedome of major adverse events (MAEs) including (1) all-cause death, (2) bowel ischemia, (3) myocardial infarction, (4) paraplegia, (5) renal failure, (6) respiratory failure, (7) stroke, and (8) Blood Loss > 1000mL at 30 Days post index procedure.
Number of subjects with Aneurysm rupture | 5 years
  The number of patients experiencing a rupture of the aneurysm will be summarized at 30 days and within each follow-up window (i.e., six months, and annually at years 1 through 5).
Number of subjects with Conversion to open surgical repair | 5 years
  The number of patients undergoing surgical conversion to open repair will be provided at 30 days and within each follow-up window (i.e., six months, and annually at years 1 through 5).
Number of subjects with Endoleak of any type | 5 years
  The number of patients with any endoleak, and patients with each endoleak type at 30 days and within each follow-up window (i.e., six months, and annually at years 1 through 5) will be summarized.
Number of subjects with Clinically significant migration | 5 years
  The number of patients with clinically significant migration will be summarized descriptively.
Number of subjects with Aneurysm enlargement | 5 years
  The number of patients with Aneurysm enlargement will be summarized descriptively. Sac enlargement is defined in the protocol as increase in late follow-up compared to the initial post-op measurement.
Number of incidence with Secondary endovascular procedures | 5 years
  The overall secondary procedure incidence and the individual component incidence will be provided.

OTHER OUTCOMES:
Number of subjects with incidence of device patency and integrity | 5 years
  Device patency and integrity will be measured by the number and proportion of patients at 30 days, 6 months, and 1 year to 5 years including Stent Kinking, Lumen Occlusion, and Stent Fracture.
Number of incidence with Distal Complications | 5 years
  The number of incidence of distal thrombosis, embolization and iliac stenosis will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Holden, MBChB, Principal Investigator — Auckland City Hospital; Michel Reijnen, MD, Principal Investigator — Rijnstate, Arnhem, the Netherlands
Locations (10):
- Germany (5):
  - Klinikum Augsburg Klinik für Gefäßchirurgie, Augsburg
  - St. Marien Hospital Bonn, Bonn
  - University Hospital Koeln, Cologne
  - University Hospital Heidelberg, Heidelberg
  - TUM Munich, Munich
- Netherlands (2):
  - Rijnstate Hospital, Arnhem
  - St Elisabeth Ziekenhuis, Dept of Vascular Surgery, Tilburg
- Auckland City Hospital, Auckland, New Zealand
- Spain (2):
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Universitario y Politécnico de La Fe, Valencia